CLINICAL TRIAL: NCT02360423
Title: A Prospective, Multi-center, Randomized Controlled Trial Evaluating the Safety and Efficacy of the CRE8 Sirolimus-Eluting Stent Versus the RESOLUTE Zotarolimus-Eluting Stent in the Treatment of Patients With De Novo Coronary Artery Lesions
Brief Title: Safety and Efficacy of the CRE8 Stent for the Treatment of De Novo Coronary Artery Lesions
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CID S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE8-China-RCT
Record Dates: First submitted 2015-02-03; First posted 2015-02-10 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CRE8 group (Experimental): CRE8 sirolimus-eluting stent system
  Interventions: Device: CRE8 sirolimus-eluting stent
- RESOLUTE group (Active Comparator): RESOLUTE zotarolimus-eluting stent system
  Interventions: Device: RESOLUTE zotarolimus-eluting stent

INTERVENTIONS:
Device: CRE8 sirolimus-eluting stent — The CRE8 stent is a flexible implantable device that can be expanded using a PTCA catheter. The stent is made of Cobalt chromium alloy and is coated with i-carbofilm.The outer surface of the stent has dedicated grooves for containing the pharmaceutical formulation, which is composed of the drug sirolimus and a mixture of long chain fatty acids.
  Arms: CRE8 group
Device: RESOLUTE zotarolimus-eluting stent — The RESOLUTE stent is a flexible implantable device that can be expanded using a PTCA catheter. The stent is made of Cobalt chromium tungsten alloy. It has been approved by CFDA in 2009 and commercially available in Chinese market
  Arms: RESOLUTE group

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy and deliverability of the CRE8 sirolimus-eluting stent and the RESOLUTE zotarolimus-eluting stent in the treatment of patients with de novo coronary artery lesions.

DETAILED DESCRIPTION:
This study consists of a randomized controlled cohort and a long stent observational cohort. The randomized controlled trial is a prospective, multi-center, non-inferior, randomized controlled trial. The control device (RESOLUTE zotarolimus-eluting stent) used in this trial was provided by Medtronic. RESOLUTE zotarolimus-eluting stent has been already approved by China Food and Drug Administration (CFDA) in 2009 and become commercially available in Chinese market. 400 patients enrolled in this trial will be randomly assigned to CRE8 group (n=200) and RESOLUTE group (n=200) in a 1:1 ratio. The long stent observational trial plans to enroll 30 consecutive patients. Patients in the observational cohort will receive the long CRE8 stent with length 38mm.All 430 patients will be required to receive clinical follow-up at 1 month, 6 months, 9 months, 12 months and annually up to 5 years after the procedure, and angiographic follow-up at 9 months after the procedure. The primary endpoint is in-stent LLL at 9 months after the procedure, and the secondary endpoints are device success rate, device-oriented cardiovascular composite endpoint, patient-oriented cardiovascular composite endpoint and stent thrombosis.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for randomized cohort:

* Age ≥18 years and ≤ 75 years, male or female without pregnancy;
* Patients with clinical evidence of asymptomatic heart disease, stable or unstable angina, or old myocardial infarction;
* De novo lesions of native coronary arteries (lesions number ≤ 2);
* Target vessel diameter between 2.25 and 4.0 mm and target lesion length ≤ 27mm by visual estimation;
* Target lesion diameter stenosis ≥ 70% by visual estimation;
* Each target lesion is permitted to implant only one stent at most, except bailout stent;
* Patients is eligible for percutaneous coronary intervention (PCI) and is an acceptable candidate for surgical revascularization (CABG);
* Patients with left ventricular ejection fraction ≥40%;
* Patients who can understand the nature of the study, agree to participate and accept angiographic and clinical follow-up, and have provided written informed consent.

Inclusion criteria for the long stent observational cohort:

* Age ≥18 years and ≤ 75 years, male or female without pregnancy;
* Patients with clinical evidence of asymptomatic heart disease, stable or unstable angina, or old myocardial infarction;
* De novo lesions of native coronary arteries (lesions number ≤ 2);
* Target lesion diameter stenosis ≥ 70% by visual estimation;
* At least one target lesion with reference vessel diameter between 2.5mm and 4.0mm and requires 38mm stent exists;
* Patients is eligible for percutaneous coronary intervention (PCI) and is an acceptable candidate for surgical revascularization (CABG);
* Patients with left ventricular ejection fraction ≥40%;
* Patients who can understand the nature of the study, agree to participate and accept angiographic and clinical follow-up, and have provided written informed consent.

Exclusion Criteria:

* Patients with acute myocardial infarction (AMI) within one week;
* Chronic total occlusion lesion (TIMI flow 0 before procedure), Left main disease and/or triple-vessel lesion that might require treatment, bifurcation lesions with a side branch diameter >2.5mm or graft lesions;
* Heavily calcified or tortuous lesions which cannot be successfully pre-dilated, and lesions which are not suitable for stent delivery and deployment;
* In-stent restenosis;
* Thrombotic lesion;
* Patients who had received any other stent in the past one year;
* Patients with acute or chronic renal dysfunction (defined as creatinine greater than 2.0 mg/dl);
* Patients with cardiogenic shock, acute infection, known bleeding or coagulation disorder, or with a history of active gastrointestinal bleeding, ulcer, cerebral hemorrhage or subarachnoid hemorrhage and stroke within 6 months;
* Patients who allergic to aspirin, clopidogrel, ticagrelor, ticlopidine, heparin, contrast agent, sirolimus, zotarolimus, polymer, Co-Cr alloy, or with contraindication to aspirin or clopidogrel or ticagrelor;
* Patients with life expectancy less than 1year;
* Patients who had participated in another investigational drug or device trial that has not completed the primary endpoint;
* Patient is in the opinion of the investigator, unable to comply with the requirements of the study protocol;
* Patients who had underwent heart transplant surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-10 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
In-stent late lumen loss (LLL) | 9months after the procedure

SECONDARY OUTCOMES:
In-stent, proximal stent edge, distal stent edge and In-segment binary restenosis rate | 9months after the procedure
In-segment late lumen loss (LLL) | 9months after the procedure
Target lesion failure (TLF) rate | 1month, 6months, 9months, 12months and annually up to 5 years follow-up
Number of participants with stent thrombosis per ARC definition | 1month, 6months, 9months, 12months and annually up to 5 years follow-up
The patient-oriented composite endpoint includes all-cause death, all MIs, or any revascularizations | 1month, 6months, 9months, 12months and annually up to 5 years follow-up
device and lesion success rates | immediately after the procedure
clinical success rate | 7 days after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Shubin Qiao, MD, Principal Investigator — Fu Wai Hospital, National Center for Cardiovasular disease
Locations (1):
- Fuwai Hospital,National Center for Cardiovasular disease, Beijing, Beijing Municipality, China